CLINICAL TRIAL: NCT03291626
Title: Postoperative Delirium: EEG Markers of Sleep and Wakefulness
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ben J.A. Palanca, Assoc Prof of Anesthesiology, Washington University School of Medicine
Other Study IDs: 201705018
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative delirium is a condition in which patients develop temporary difficulties in maintaining attention and thinking clearly. These new problems can appear after surgery and change throughout the day. This confusion can last several days.

The overall purpose of this study is to measure brain activity during sleep and wakefulness to learn about their relationships to delirium after surgery. While participants may not feel like their normal self during the study, they are in the best position to help us learn how to improve the recovery of brain function and sleep in others having surgery. The investigators need to learn from those who have and have not become confused after their surgical procedure.

DETAILED DESCRIPTION:
Postoperative delirium is a condition that can develop in some older patients after they have surgery and receive general anesthesia. Patients that develop delirium have difficulty maintaining attention and thinking clearly. Both of these issues can come and go throughout the day. The incidence of postoperative delirium is greater than 25% and is associated with longer hospitalization and increased risk of persistent mental and physical decline. It is thought that this disorder may be preventable, but there is no agreed upon way of identifying which patients are at risk for delirium prior to their surgery. Additionally, patients with atypical delirium are often misdiagnosed or undiagnosed postoperatively.

Based on previous research, the researchers have hypothesized that delirium may be directly related to wakefulness and sleep problems, as shown on electroencephalography [EEG]. EEG is a test that records the electrical activity of brain through placement of small wires on a person's scalp. In light of this, the purpose of this study is to evaluate sleep and wakefulness using EEG before, during and after surgery in order to discover any abnormalities of sleep or wakefulness that associate with postoperative delirium onset, severity, and length of recovery. Subjects in this study will have preoperative at home sleep testing performed, using a device called the Sleep Profiler, and questionnaires administered to characterize their mental function and brain function prior to surgery. When they arrive for their scheduled surgery, the subjects will be fitted with the Sleep Profiler to record brain activity during surgery and after surgery for 5 days. Postoperatively, the subjects will be asked to do simple tasks like move toes and fingers and to answer questions that assess their mental state.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Age 60 or older
3. Scheduled for cardiac surgery requiring cardiopulmonary bypass for coronary artery bypass grafting and/or heart valve repair/replacement

Exclusion Criteria:

1. Pre-existing delirium or dementia
2. Legal blindness or severe deafness
3. Surgery requiring deep hypothermic circulatory rest

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants recruited from the Barnes Jewish Hospital in St. Louis receiving elective cardiac or major thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Change from pre-operative awake EEG measurement to sleep EEG measurement | Record at baseline visit or, if the subject is an inpatient, once during the day compared to record obtained overnight either at home or in the hospital
  Awake EEG recorded at baseline, sleep EEG using Sleep Profiler
Change in baseline diagnosis of delirium to hospital discharge | Diagnosis at baseline, then diagnosis change evaluated 2 times daily post-operatively until hospital discharge or post-operative day 5, whichever occurs first.
  Delirium diagnosed using the validated instrument Confusion Assessment Method, Long Form

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD, PhD, Principal Investigator — Washington University in St Louis SOM
Locations (1):
- Barnes-Jewish Hospital/Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with the National Sleep Research Resource within three years after completion of the study. We will register our observational study on clinicaltrials.gov and publish a protocol of our approach and pre-specified analyses by the end of Year 2 of funding.
Supporting Information: Study Protocol
Time Frame: Data will be made available within 3 years of study completion and publication and will be available indefinitely.
Access Criteria: Permission from the principal investigator is required for access.
URL: https://sleepdata.org/

REFERENCES:
- [Derived] Luong AH, Smith SK, Bhatia K, Kafashan M, Nguyen T, Hyche O, Schill M, Damiano RJ Jr, Palanca BJA. New-Onset Postoperative Atrial Fibrillation and Preoperative Sleep in Cardiac Surgical Patients. Ann Thorac Surg Short Rep. 2024 Jul 26;3(1):258-263. doi: 10.1016/j.atssr.2024.07.010. eCollection 2025 Mar. PMID 40098862
- [Derived] Smith SK, Nguyen T, Labonte AK, Kafashan M, Hyche O, Guay CS, Wilson E, Chan CW, Luong A, Hickman LB, Fritz BA, Emmert D, Graetz TJ, Melby SJ, Lucey BP, Ju YS, Wildes TS, Avidan MS, Palanca BJA. Protocol for the Prognosticating Delirium Recovery Outcomes Using Wakefulness and Sleep Electroencephalography (P-DROWS-E) study: a prospective observational study of delirium in elderly cardiac surgical patients. BMJ Open. 2020 Dec 13;10(12):e044295. doi: 10.1136/bmjopen-2020-044295. PMID 33318123